CLINICAL TRIAL: NCT03115827
Title: Norepinephrine-targeted Therapy for Action Control in Parkinson Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: H. Lundbeck A/S (Industry); American Academy of Neurology (Other)
Responsible Party: Principal Investigator, Katherine Eder McDonell, Assistant Professor of Neurology, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VUMC54580
Record Dates: First submitted 2017-03-09; First posted 2017-04-14 (Actual); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Droxidopa; Carbidopa

STUDY DESIGN:
Intervention Model Description: This is a single-arm study enrolling 15 patients that will all receive the experimental treatment.
Masking Description: All patients will receive the same treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): Droxidopa 600mg by mouth twice a day and carbidopa 200mg by mouth twice a day for 4 weeks
  Interventions: Drug: Droxidopa; Drug: Carbidopa

INTERVENTIONS:
Drug: Droxidopa — Droxidopa will be started at 100mg twice a day and titrated up to a maximum of 600mg twice a day
Drug: Carbidopa — Carbidopa 200mg twice a day

SUMMARY:
The purpose of this study is to find out whether droxidopa, a medication that increases norepinephrine levels, may be effective in improving some aspects of cognition and movement in Parkinson's disease (PD).

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a progressive neurodegenerative disorder that affects 1 million people in the United States. PD causes a variety of disabling symptoms, which impact movement as well as cognition. Historically, we have relied on medications that increase dopamine levels to treat PD, although we are recognizing more and more that other chemicals in the brain are involved in PD as well.

Droxidopa (Northera) is an approved drug for the treatment of low blood pressure in PD. It is a norepinephrine precursor, which is converted in the body to the neurotransmitter norepinephrine. This is a chemical that the body normally makes that has a variety of important activities in the brain and peripheral nervous system. In PD, the cells that make norepinephrine die off as part of the disease process. Therefore, people with PD often have low levels of norepinephrine in their blood and in their spinal fluid. Norepinephrine is important for maintaining blood pressure, which may be one reason that some people with PD have problems with their blood pressure falling too low when they stand up. This can lead to symptoms such as dizziness, lightheadedness, feeling faint, or sometimes passing out.

Droxidopa has been approved by the FDA for the treatment of low blood pressure in Parkinson's disease. However, as norepinephrine is also important for a lot of processes that happen in the brain as well, we believe that this medication may be also helpful for some of the other symptoms of PD. In particular, norepinephrine plays a key role in brain networks that are important for attention, decision making, and controlling movements and actions. In order for norepinephrine to reach the brain, it must cross the blood-brain barrier. Therefore, in this study we will be giving droxidopa along with carbidopa, which stops your body from breaking down norepinephrine in the blood stream and allows it to get into the brain. This is a medication that is often given in Parkinson's disease along with levodopa in the form of carbidopa-levodopa, or Sinemet. This medication works the same way with levodopa in helping it get into the brain and improve the symptoms of PD. The only difference is that levodopa works like the chemical dopamine, whereas droxidopa works like norepinephrine. Up to this point, we have not had a way to correct the low norepinephrine levels in Parkinson's disease. Therefore, this study gives us the chance to investigate the effectiveness of a potential new treatment for PD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Nondemented man or woman 18 years of age or older with idiopathic PD based on the UK Parkinson Disease Society Brain Bank Clinical Diagnostic Criteria (refer to Appendix C for the criteria)
2. Unified Parkinson Disease Rating Scale (UPDRS) motor scores OFF medication consistent with postural instability gait difficulty (PIGD) subtype
3. Symptoms of freezing or falls
4. Able to walk at least 10 meters
5. Medically stable outpatient, based on the investigator's judgment
6. The patient must be willing and able to give written informed consent prior to performing any study procedures.

Exclusion Criteria:

1. Score of 21 or lower on Montreal Cognitive Assessment
2. Sustained supine hypertension greater than or equal to 180 mmHg systolic or 110 mmHg diastolic, or have these measurements at their Baseline Visit (Visit 2). Sustained is defined as measurements persistently greater at 2 separate measurements at least 10 minutes apart with the subject supine and at rest for at least 5 minutes.
3. Concomitant use of vasoconstricting agents such as ephedrine, dihydroergotamine, or midodrine. Concomitant use of other noradrenergic medications, such as serotonin-norepinephrine reuptake inhibitors (SNRI's) is also contraindicated. Patients must stop taking these drugs at least 2 days or 5 half-lives (whichever is longer) prior to their baseline visit and throughout the duration of the study.
4. Diagnosis of hypertension that requires treatment with antihypertensive medications (short-acting antihypertensives to treat nocturnal supine hypertension are allowed in this study)
5. Women of childbearing potential
6. Any significant uncontrolled cardiac arrhythmia
7. History of myocardial infarction, within the past 2 years
8. Current unstable angina
9. Congestive heart failure (NYHA Class 3 or 4)
10. History of cancer within the past 2 years other than a successfully treated, non-metastatic cutaneous squamous cell or basal cell carcinoma or cervical cancer in situ
11. History of stroke
12. Gastrointestinal condition that may affect the absorption of study drug (e.g., ulcerative colitis, gastric bypass)
13. Musculoskeletal disorders such as severe arthritis, post knee surgery, hip surgery, or any other condition that the investigators determine may impair assessment of gait
14. History of myocardial infarction, uncontrolled cardiac arrhythmia, unstable angina, congestive heart failure, or stroke
15. Untreated closed angle glaucoma
16. Musculoskeletal or other disorders that may impair assessment of gait
17. Any major surgical procedure within 30 days prior to the Baseline visit
18. Previously treated with droxidopa within 30 days prior to the Baseline visit
19. Currently receiving any other investigational drug or have received an investigational drug within 60 days prior to the Baseline visit
20. Known or suspected alcohol or substance abuse within the past 12 months (DSM-IV definition of alcohol or substance abuse)
21. Any condition or laboratory test result, which in the Investigator's judgment, might result in an increased risk to the patient, or would affect their participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine McDonell, MD, Principal Investigator — Vanderbilt Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1
Started | 15
Completed | 12
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Develop an Adverse Event During the 7-week Treatment Period That is Determined to be Likely Related to the Study Medications.
Description: Safety will be defined by the percent of subjects who develop an adverse event during the 7-week treatment period that is determined to be likely related to the study medications.
Time Frame: 7 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1
Number analyzed (Participants) | 15
Participants | 8

2. Primary Outcome: Number of Participants Who Discontinue the Study Drug Due to Adverse Effects During the 7-week Treatment Period.
Description: Tolerability will be defined by the number of patients who discontinue the study drug due to adverse effects.
Time Frame: 7 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1
Number analyzed (Participants) | 15
Participants
  Participants that discontinued due to SAEs | 2
  Participants that discontinued due to mild AEs | 1
  Participants that did not discontinue | 12

3. Secondary Outcome: Maximum Tolerated Dose
Description: The mean maximum tolerated dose of droxidopa reached by the study participants
Time Frame: Week 4 to Week 7
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Arm 1
Number analyzed (Participants) | 15
mg/day | 1053 (267)

4. Secondary Outcome: Percent Compliance
Description: Percent compliance is defined as the percent of study participants who take greater than or equal to 70% of the assigned dosage
Time Frame: 7 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1
Number analyzed (Participants) | 15
Participants | 11

5. Secondary Outcome: Change in Stop-Signal Reaction Time From Baseline to Week 7
Description: The Stop-Signal reaction time is a computerized test that assesses reaction time and response inhibition
Time Frame: baseline and week 7
Measure: Mean (Standard Deviation); unit: change in SSRT in seconds
Arm/Group | Arm 1
Number analyzed (Participants) | 15
change in SSRT in seconds | -14.38 (40.42)
Statistical Analysis 1: Comparison: Arm 1; Test type: Other; p = 0.6, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 11 weeks
Description: The definitions used to collect the adverse event information does not differ from the clinicaltrials.gov definitions. Serious adverse event information was collected over the phone at the time of onset. Adverse Event information was collected at each study visit including baseline, visit 1, visit 2, visit 3, and the follow-up visit.
Arm/Group | Arm 1
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 10/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=15)
transient cholecystitis (Gastrointestinal disorders) | 1 (1)
ventral hernia (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=15)
Nausea (Gastrointestinal disorders) | 2 (2)
Dry Mouth (General disorders) | 1 (1)
Increased Freezing (Nervous system disorders) | 1 (1)
Conjunctival Hemhorrage (Eye disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Brief Confusional Episode (Psychiatric disorders) | 1 (1)
Influenza-like symptoms (General disorders) | 1 (1)
Increased Uncoordinated Movements (Nervous system disorders) | 1 (1)
Increased Foot Dystonia (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was an open-label, dose-titration, safety and tolerability pilot study with a small sample size (n=15). Additionally, there was no placebo arm or comparison group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-31): https://cdn.clinicaltrials.gov/large-docs/27/NCT03115827/Prot_SAP_000.pdf